Family Model of Diabetes Self-Management Education in Faith Based Organizations in the Republic of the Marshall Islands Study Title:

PI (researcher): Sheldon Riklon, MD

# FAMILY MODEL DIABETES SELF-MANAGEMENT AND EDUCATION IN FATIH BASED ORGANIZATIONS IN THE REPUBLIC OF THE MARSHALL ISLANDS

NCT05502016

V.9; 10/4/2024


Organizations in the Republic of the Marshall Islands

PI (researcher): Sheldon Riklon, MD

# KEY INFORMATION FOR FAMILY MODEL OF DIABETES SELF-MANAGEMENT EDUCATION (DSME) IN FAITH BASED ORGANIZATIONS:

MELELE KO RAORŌK KŌN EKKATAK EO NAETAN "FAMILY MODEL OF DIABETES SELF-MANAGEMENT EDUCATION (DSME)" IM REJ KOMMAN ILO DOULUL KO AN KABUÑ:

We are asking you to choose whether or not to volunteer for a research study about helping persons with diabetes and their family members learn how to manage diabetes. Classes for this study will be done in a church or other faith-based setting.

Kōmij kajjitōk bwe kwōn kelet elañe kwōj kōnaan ak jab kōnaan bōk konaam ilo ekkatak in ñan jibañ armij ro ewōr aer nañinmej in tōñal koba baamle ko aer ñan katak kōn nañinmej in tōñal im wāwein ko ñan kōjparok. Kilaaj ko an ekkatak in renaj kōmman ilo imōn jar ko ak jikin ko jet an mwōn jar ko.

This page gives you key information to help you decide whether to participate. We have included detailed information after this page. Ask the research team questions. If you have questions later, the contact information for the research investigator in charge of the study is below.

Pepa in ej kwalok melele ko raurōk nan jiban iok komman kelet eo am im kalikar kwoj ke bok konaam. Emoj droor melele ko remelijlok ālikin pepa in. Lelok kajjitōk ko am nan team eo ej bok eddoin ekkatak in. Elane ewor am kajjitōk tok ālik, melele ko nan tobar rijerbal ro an ekkatak in rej bed āliktata in pepa kein.

# WHAT IS THE STUDY ABOUT AND HOW LONG WILL IT LAST? EKKATAK IN EJ KŌN TA IM EWI AITOKAN?

By doing this study, we hope to see whether Marshallese patients with diabetes can improve their health and quality of life if they and their families learn together about managing their diabetes. We also want to learn if teaching about diabetes in a church setting is better than teaching in other places. To test this, we will measure if their diabetes improves. Up to 288 Marshallese adults (ages 18 years and older) with diabetes and one to two of their family members may be part of this study. Your participation in this research will last about 10-12 months with approximately 10 hours of diabetes education over an 8-12 week period and you will participate in three to five data collection events. If you join the study, you will be asked to attend diabetes management classes and data collection sessions where we collect health information. You may be asked to participate in an interview and short survey to talk about how well the classes worked for you and the educators' ability to teach the classes.

Ilo ad kōmmane ekkatak in, jej kōjatdikdik ke jenej maroñ loe elañe Rimajōl ro ewōr aer nañinmej in tōñal remaroñ kōkmanman lok ājmour ko aer im jokkin mour ko aer elañe er im baamle ko aer renej ekkatak ibben dron kōn bōbrae nañinmej in tōñal ko aer. Jej bar kōnan jelā elañe katakin kōn nañinmej in tōñal ilo mwōn jar ko emman lok jen jikin ko jet. Ñan kajjioñ men in, jenej etale elañe nañinmej in tōñal ko aer rej emman lok. Ewōr 288 rutto in Majōl ro (18 iiō im rutto lok) im ewōr aer nañinmej in tōñal im 1-2 uwaan baamle ko aer renej maroñ mōttan ekkatak in. Ilo am bōk konaam ilo ekkatak in eo aitokan enej tarrin 10 ñan 12 allōñ koba tarrin

Organizations in the Republic of the Marshall Islands

PI (researcher): Sheldon Riklon, MD

10 awa in ekkatak kōn nañinmej in tōnal ilo 8-12-wiik aitokan im konej bar bōk konaam ilo jillu nan emen ien ko nan ebbōk melele ko am. Ne konej kobatok ilo ekkatak in, renej kajjitōk ibbam nan bed ilo kilaaj in kejbarok nañinmej in tōnal im ien bōk am ae melele ko am ikijjien ejmour. Remaron kajjitōk ippam bwe kwōn bōk kunaam ilo juon iien bok melele im kajitōkin eok kōn ewi jonan an emman an kilaaj ko jerbal nan kwe im ewi jonan an rūkaki eo jeļā kilen katakin kilaaj ko.

#### WHY MIGHT I CHOOSE TO VOLUNTEER FOR THIS STUDY?

#### ETKE INEJ MAROÑ KELET BWE IN BŌK KONAŌ ILO EKKATAK IN?

You are being invited to join in this study because you either have diabetes or because a family member with diabetes has invited you to join with them. As a person in the study, you will attend diabetes education classes led by a trained diabetes teacher. During these classes you will learn about healthy eating, being active, tracking blood sugar, and other skills that help people to manage diabetes. Being in the study may help your health improve and may help other persons with diabetes in the future. For a complete description of benefits, refer to the Full Consent.

Emōj kajjitōk ibbam nan koba tok ilo ekkatak in konke ewor am naninmej in tonal ak konke juon eo uwaan baamle eo am ewor an naninmej in tonal ej kur tok eok nan koba tok ibbeir. Einwot juon eo ej bed ilo ekkatak in, konej bed ilo kilaaj in tonal kein im rej komman jen juon eo ewor an kapeel ikkijen katakin kon naninmej in tonal. Ilo ien kilaaj kein kwonej ekkatak kon kejbarok ad mona, makutkut, etale tonal eo am, im kapeel ko jet im rej jiban armej bobrae naninmej in tonal. Am bed ilo ekkatak in emaron jiban bwe kwon ajmour lok, im emaron jiban armij ro ewor aer naninmij in tonal iliju im jeklaj. Nan melele ko remelijlok ikijien emman ko an ekkatak in, kwonaj riiti pepa in Full Consent eo elikin pepa in.

#### WHY MIGHT I CHOOSE NOT TO VOLUNTEER FOR THIS STUDY?

# ETKE INEJ KELET BWE IN JAB BŌK KONAŌ ILO EKKATAK IN?

There is the chance that someone could find out about your private health information, but we will take special care to reduce this risk. By taking part in the educational sessions other people in the session may learn information about you if you talk about yourself.

Emaron wor ien eo im juon armij emaron jela kon melele ko ikijen ajmour eo am, botaap jenaj kojparok bwe en jab walok wawein in. Ilo am bok kilaaj ko, armij ro jet remaron jela melele ko kon kwe make elane kwonaj kenono kaki.

There is no guarantee that the study will help you. For a complete description of risks, refer to the full Consent.

Ejjelok kallimur ke ekkatak in enaj jibañ eok. Nan melele ko remelijlok ikijien emman ko an ekkatak in, kwonaj riiti tarlepen pepa in Mālim (Consent) eo ālikin pepa in.

Organizations in the Republic of the Marshall Islands

PI (researcher): Sheldon Riklon, MD

#### DO I HAVE TO TAKE PART IN THE STUDY?

#### IJ KE AIKUJ BŌK KONAŌ ILO EKKATAK IN?

No. It is okay to say no. If you decide to take part in the study, it should be because you really want to volunteer. You will not lose any services, benefits, or rights you would normally have if you choose not to volunteer.

Jaab. Ejjelok bwōd ne kwonaj ba jaab. Elane kwonaj erra in bōk konaam ilo ekkatak in, ej aikuj kōnke kwe make kwōj kōnaan bōk konaam. Eban jako jabdrewōt maron ko am ak jiban ko ekka am būki elane kwonaj kelet in jab bōk konaam.

# **University of Arkansas for Medical Sciences Informed Consent Form**

If you want to know more about the research, let the study team know so they can give you more information. You can reach the local research team at 692-456-4875. You can also send an email to <a href="wibing@uams.edu">wibing@uams.edu</a>.

Eļanē kwoj koņaan jeļā eļapļok kon ekkatak in, kojeļā ik team in ekkatak eo bwe ren maronē lewaj eļapļok meļeļe ko. Kwomaronē topar team in ekkatak eo ijin ilo 692-456-4875. Kwomaronē bar jilkinļok juon email nan wibing@uams.edu

Also tell the study team if you have decided you don't want to be in the study. It is perfectly okay to say no.

Kwōn bar kōjeļāik team in ekkatak eo eļanē emōj am kelet bwe kwōn jab pād ilo ekkatak eo. Ejjelok jorrāān ne kwoba jaab.

- We are asking you to be in a research study. You do not have to join the study. Jej kajitōk ibbam bwe kwōn bed ilo ekkatak in. kwojjab aikuj bed elañe kwojjab kōnan.
- Please take as much time as you need to read this form and decide what is right for you. Jouj im bok am ien nan riiti pepa in im kelet ta eo emman nan kwe.

#### Why am I being asked to be in this research study?

#### Etke rej kajjitōk ibba bwe in bed ilo ekkatak in?

• We want to learn more about teaching about diabetes self-management. Jej konan katak elap lok kon katakin kojebarok naninmej in tonal

Organizations in the Republic of the Marshall Islands

PI (researcher): Sheldon Riklon, MD

 This study will help us learn more about whether Marshallese patients with diabetes can improve their health and quality of life if they and their family learn about managing their diabetes in a church setting.

Ekkatak in enej jibañ kōj jelā elaplok melele ko elañe rimajōl ro ewōr aer nañinmej in tōñal im remaroñ kōkmanmanlok ājmour ko aer im wāwein jokkunmour ko aer elañe er im baamle ko aer renej ekkatak wāwein kōjebarok nañinmej in tōñal ko aer ilo mwōn jar ko.

• We are asking people like you who have diabetes or have been invited by a family member with diabetes to help us.

Kōmij kajjitōk ibben armej einwōt kwe eo im ewōr an nañinmej in tōnal ak juon eo emōj kūr tok eok jen juon ian ro nukum im ewōr an nañinmej in tōnal nan jiban kōm.

 Up to 240 Marshallese adults (ages 18 years and older) with diabetes and one to two of their family members may be part of this study.

Ewōr 240 rutto in Majōl ro (18 iiō im rutto lok) im ewōr aer nañinmej in tōnal im juon ian baamle ko aer bwe ren bar mōttan ekkatak in.

# What if I don't understand something?

### Elañe ewōr jabdrewōt men eo ijjab melele kake?

- This form may have words you don't understand. If you'd like, research staff will read it with you. Emaron wor melele ko kwojjab melele kaki ilo pepa in. Elane kwoj konaan, ro rej jerbal ilo ekkatak in remaron riiti im etale pepa in ibbam
- You are free to ask questions at any time before, during, or after you are in the study. Kwomaron komman am kajitok jabdrewot ien mokta, ien eo, ak ālikin ekkatak in.
- Please ask as many questions as you like before you decide whether you want to be in this study. Jouj im letok aolep am kajjitōk mokta jen am kelet elañe kwoj kōnan bed ilo ekkatak in.

### What will happen if I say yes, I want to be in this study?

### Ta enej walok elañe inaj ba aet, ij kōnan bed ilo ekkatak in?

We first will see if you qualify to be in the study. We will ask if you...

Jenaaj lale mokta elane kwoj ekkar nan bed ilo ekkatak in. Jenaj kajjitok ibbam elane kwe...

Identify as Marshallese, juon ri Majol

Organizations in the Republic of the Marshall Islands

PI (researcher): Sheldon Riklon, MD

• Are 18 years or older. 18 am iiō ak rutto lok.

- Have type 2 diabetes (HbA1c equal or greater than 6.5) or are a family member of a person with type 2 diabetes. ewor naninmij in tonal taip 2 ibbam, ak juon eo uwaan baamle eo am ewor an naninmej in tonal taip 2 (HbA1c eo ej einwot ak laplok jen 6.5).
- Have received DSME in the past five years. emōj am bōk kilaaj in DSME ilowaan iiō ko lalem rej mootlok.
- Have at least one family member who will agree to take part in the study with you. ewor juon armij uwaan baamle eo am im emoj an errā in bok konaan ilo ekkatak in ibbam.
- Plan to move out of the area in the next 12 months Kwōj lōmnak in emmakit jen jikin ko rej kōmmane ekkatak eo je ilowaan 12 allōn ko.
- Have an illness that would prevent you from fully participating in the classes such as terminal illness, non-ambulatory, severe mental illness, severely impaired vision or hearing, or eating disorder Ewōr am nañinmej ko renej bōbraik eok jen am bed ilo kilaaj ko einwōt nañinmej ko ejjelok unokaer ak rejjab maroñ kōmadmōdi, jab maroñ jutak make ian ak ejjab maroñ etetal, nañinmej in kōmālij, jab lolok ijen ak jaroñroñ, ak ejjab jejjet wāwein aer mōñā.

If you qualify, we will do these things:

## Elañe ekkar nan bok konaam, kom naj kommani wawein kein:

Enroll you in diabetes education classes. Classes will cover approximately 10 hours of diabetes education over an 8-12 week period, and each class will last between 60 and 90 minutes. Classes for this study will be done in a church or other faith-based setting. Participants and family members will attend classes in a group setting with other participants and their family members. If you agree to be contacted via text message, we will text you each week during classes to remind you of the date, time, and location of your class. We may also text you to remind you of upcoming data collection events. During these classes you will learn about healthy eating, being active, tracking blood sugar, and other skills that help people to manage diabetes. The family members you invite will be asked to join the study and participate in diabetes education classes. Family members can attend the classes, even if they are not in the study. Kadeloñ etam ilo kilaaj in nañinmij in tōnal ko. Kilaaj ko ikijien nañinmej in tonal renaaj tarrin 10 awa aitokier ilowaan 8-12 wiik. Im kajojo iien kilaaj kein enaj 60 nan 90 minit aitokier. Kilaaj ko renaj kōmman ilo mwōn jar ko ak bar juōn jikin an mwōn jar ko. Ro rej bōk konaer im uwaan baamle ko aer renej bed ilo kilaaj kein ilo juon doulul in armej ibben ro jet mõttan ekkatak in im ro uwaan baamle ko aer. Ne kwonej errā bwe jen tōbar eok ilo text message ak jeje waj ilo cellphone eo am, jenej jeje waj ilo kajojo wiik nan kakemejmej eok kon ien eo, awa eo, im ia eo kilaaj eo enej komman. Ilo kilaaj kein, kwonaj ekkatak kōn wãwein kōjebarok am mōnā, makūtkūt im exercise, etale jonan tōnal, im wāwein ko jet remaron jiban ikijien naninmej in tonal. Jenaj bar kajjitok ibben armij ro nukum kwar kūr er bwe ren bar bōk konaer ilo kilaaj ko ikijien nañinmij in tōnal. Armij ro nukum remaron bed ilo kilaaj ko, jekdron ne raar jab lelok etaer nan ekkatak in.

Organizations in the Republic of the Marshall Islands

PI (researcher): Sheldon Riklon, MD

Ask about demographic information such as your name, address, phone number, date of birth, sex, marital status, number of persons in your home, education, employment, race/ethnicity, health behavior, understanding, and health care access. Ask about information related to your health such as height, weight, pregnancy status, tests for diabetes, blood pressure, support from your family, managing your weight, exercise, what medications you take, what you eat and drink and what size shoe you wear. Kem naaj kajjitōk kōn meļeļe ko an juon jarlepju in armej (demographic information) āinwōt etam, atōrej in jikin jokwe, talboon nōmba, raan in ļotak, kōrā ke emmaan, rimare ke jaab, oran armej ilo mweo mwōm, jikuul, jerbal, jen aelōn ta/kurub in armej ta, mwil ko rejelōt ājmour, jeļā im meļeļe, kab maron taktō. Kem naaj kajjitōk kōn meļeļe ko ikijjien ājmour me am āinwōt jonan aetok, eddo, bōroro, kakolkol in naninmej in tonal ko, aebūļat, jiban jen baamle eo am, kojparok eddo eo emman, exercise im makūtkūt, uno ko kwoj būki, monā ta ko kwoj kani im dan ta ko nimom im jaij ta juuj kwoj konake.

- Ask if you would like to join a UAMS Facebook group providing continued education, reminders for upcoming education or data collection events, and connecting you with others who participate in this research study for support. Participation in the Facebook group is completely voluntary. You may still participate in the research study even if you chose not to participate in the Facebook group. Kajjitōk ne kwōj kōṇaan kobaļok ippān juon an UAMS Facebook group im ej kōṇṇaan katak, kakememej ko kōn ien kilaaj ko ak ien kakōlkōl ko, im kobaik ro rej bōk kwoṇaer ilo ekkatak in nan jipan eok. Aṃ bōk kwoṇaaṃ ilo Facebook group in ej aṃ wōt pepe. Kwōj maron wōt bōk kwoṇaaṃ ilo ekkatak in mene kwōj kālet in jab bōk kwoṇaaṃ ilo Facebook group eo.
- Bilingual staff members will read the questions out loud and fill out the form with you, if like. You don't have to answer any questions you don't want to answer. Rijerbal ro rej kajin majōl renaj riiti kajjitōk ko im kanne pepa in ibbam, ñe kwōj kōnaan. Kwōjjab aikuj uwaak jabdewōt kajjitōk elañe kwojjab kōnaan
- Each church will be assigned to one of two groups. Churches in one group will begin classes immediately after the first data collection event. Churches in the second group will have the same classes but they will start later than the classes for the first group. Kajojo mwōn jar ko renaj maroñ bed ilo juon ian doulul ko ruo. Mwōn jar ko ilo doulul eo juōn renaj mōkaj im jino kilaaj ko aer ālikin wōt aer ebbōk melele ko aer. Mwōn jar ko ilo doulul eo kein karuo renej bōk ejja kilaaj ko wōt bōtaab renaj jino ālikin doulul eo juōn.
- Before classes begin, after classes end, and at 4 months after the classes, we will collect information from you and your participating family members. We may also collect information from you 12 months after classes. These data collection events will include measuring your height, weight, and blood pressure. You and any participating family members will also have some tests done to track blood sugar over time. This test will require a finger prick to get a small drop of blood. At two to three of the data collection events, you and any participating family members will also fill out surveys that ask questions about diabetes care and management. Each of the 3-5 study visits will last

Organizations in the Republic of the Marshall Islands

PI (researcher): Sheldon Riklon, MD

about 2-4 hours. Jenaj ebbōk melele (data collection) jen kwe im ro nukum raar errā in bōk konaer ilo ien kein: mokta jen an jino kilaaj kein, ālikin an jemlok kilaaj eo eliktata, im 4 allōn ālikin kilaaj kein. Kem maron bar ebbōk meļeļe ko jen kwe 12 allōn ālikin kilaaj ko. Melele ko jenaj aini ilo ien data collection ko renaj einwōt kein: jonan aitokam, eddoūm, im blood pressure ak aibōlat. Kwe im ro nukum rej bed ilo ekkatak in naj bar lale jonan tōnal ko aer. Kakōlkōl kein renaj aikuj bwe jen wākār jabon adiin peim im bōk jidrik bōtōktōk. Ilo ruo lak nān jilu iaan iien data collection kein, kwe im eo uwaan baamle eo am naaj bareinwōt kanne survey ko rej kajjitōk kōn naninmij in tōnal im wāwein kōjbaroke. Ilo kajojo ien data collection kein 3-5, renaj bōk tarrin 2-4 awa aitokier.

## How long will this study take?

#### Ewi aitokan ekkatak in?

If you agree to join this study, you will participate in approximately 10 hours of diabetes education over an 8-12 week period and you will participate in three to five data collection events. The entire study including, the diabetes education classes and data collection will be over a period of about twelve-months. Eļanīne kwōj errā in kobaļok ilo ekkatak in, kwōnaaj bōk kuṇaaṃ ilo tarrin10 awa kilaaj in nanīnmej in tōnāl iuṃwin 8 nān 12 wiik im kwōnaaj bar bōk kuṇaaṃ ilo jilu nān ļalem iien ebbōk meļeļe ak kakolkol ko. Aolepen ekkatak in ekoba, kilaaj in ekkatak kōn nanīnmej in tōnāl ko im iien ebbōk meļeļe im renaaj kōṇṇṇan iuṃwin tarin jonoul ruo-allōn.

#### What if I say no, I do not want to be in this study?

# Ak ne inaj ba jaab, ijjab konaan bed ilo ekkatak in?

Nothing bad will happen. Ejjelok jorāān enaj walok.

## What happens if I say yes, but change my mind later?

#### Ta enaj walok elaññe in aba aet, innem oktak aō lemnak tokelik?

- You can stop being in the study at any time. Komaron bojrak jen ekkatak in jabdewot ien.
- Nothing bad will happen. Ejjelok jorāān enaj walok.
- If you decide to stop being in the study, call Dr. Sheldon Riklon at (479)-713-8658. You can also call 692-456-4875 and speak with a member of the local research team in the Marshall Islands. Elañe kwōj lōmnak in bōjrak jen ekkatak in, call e Dr. Sheldon Riklon ilo (479)-713-8658. Kwomaroñ bar kūrļok 692-456-4875 im kenono ippān juon uwaan team in ekkatak eo ijin ilo Majōļ in.


Organizations in the Republic of the Marshall Islands

PI (researcher): Sheldon Riklon, MD

## Will it cost me anything to be in the study?

#### Ewor ke onāān ao bed ilo ekkatak in?

The study will not cost you anything. Ejelok oneen am bok konaam ilo ekkatak in.

# Will I be paid for being in the study?

## Enaaj ke wor ao kolla kon ao bok konao ilo ekkatak in?

Yes. We will give you \$20 to thank you for your time each time we collect information from you. You will not be paid to attend the educational classes. If you complete all three to four data collection events, you will receive \$60 to \$80. You will only receive the incentive for the times you attend the events. Persons who attend all of the educational sessions will receive an additional \$20. If you attend all three or four data collection events and all the classes, you will receive a total of \$80 to \$100. If you are asked to participate in a qualitative interview and short survey, you will receive an additional \$20. We may hold an additional data collection event 12 months after classes. You will be paid an additional \$20 for participating in that data collection event. Aet. Kem naaj lewaj \$20 tala nan kammoolol eok kon iien ko am ilo kajjojo iien kemij ebbōk meļeļe jen ippam. Kem ban koļļāik eok ikijjien am pād ilo kilaaj in katak ko. Eļanne emōj am kadedeikilok aolep iien ebbōk melele ko jilu nan emān, kem naaj lewaj \$60 nan \$80. Kwōnaaj bōk wōt kein kammoolol ko kōn iien ko kwōj pād ilo iien ebbōk melele ko. Armej ro rej pād ilo aolep kilaaj ko enaaj bar etal nan er juon \$20. Eļanne kwoj pād ilo aolep iien ebbok meļeļe ko jilu nan emān im aolep kilaaj ko, enaaj iwoj jonan in \$80 nan \$100. Eļanne kem naaj kajjitōk bwe kwōn bōk kuṇaam ilo juon iien kajjitokin eok im bok melele, enaaj iwōj juon am bar \$20. Kem maron bar kommane juon iien ebbok melele 12 allon alikin kilaaj ko. Kem naaj kölläiki eok bar juon \$20 kön am bök kunaam ilo iien ebbök melele ne.

#### Will being in this study help me in any way?

#### Ekkatak in enaj ke jiban na ilo jabdewot wawein?

Being in the study may or may not help you but may help people manage their Type 2 Diabetes in the future. What we learn may help you in the following ways: Am pād ilo ekkatak in emaroā ak emaroā jab jipaā eok bōtaab emaroā jipaā armej ro lale im kōjparok naāinmej in Taip 2 tōāal ko aer ilju im jekļaj. Jemlok in ekkatak in emaron jipaā eok ilo wāwein kein rej ellaajrak:

 You may learn how to better manage Type 2 Diabetes Kwomaron katak wawein eo emmanlok nan lale im kojparok naninmej in Taip 2 Tonal


Organizations in the Republic of the Marshall Islands

PI (researcher): Sheldon Riklon, MD

 You may learn how to better support your family members who have Type 2 Diabetes Kwomaron katak wawein eo emmanlok nan jiban ro uwaan baamle eo am im ewor aer naninmej in Taip 2 Tonal

## What are the risks of being in this study?

## Ta kauwōtata ko remaron walok jen ao bed ilo ekkatak in?

The risks are:

#### Kauwotata ko rej:

- The risks for this study are no more than what happens in everyday life. Kauwotata ko ekkā aer walok jen raan nan raan.
- You may experience discomfort from the finger prick. Komaron abonono ilo aer wākāre addin bweūm.
- Someone could find out that you were in the study and learn something about you that you did not want others to know. We will do our best to protect your privacy, as explained in more detail later in this form. Ro jet remaron jelā ke kwoj bed ilo ekkatak in im jelā melele ko am im kwojjab konan bwe ro jet ren jelā. Jenaj kajjion jonan wot am maron kojebarok melele ko am, einwot an komeleleik elap lok ijiko tok imaan ilo pepa in
- By taking part in the educational sessions other people in the session may learn information about you if you talk about yourself. Ilo am naj bed ilo kilaaj ko, armij ro jet ilo kilaaj eo remaroñ roñ melele ko am elañe konaaj kenono kôn kwe make.

#### What if I get sick or hurt while I'm in this study?

#### Elane inaaj naninmej ak joraan ilo ao bed ilo ekkatak in?

If you get hurt when you are here for the study, we will help you get the care you need. This may include first aid, emergency care, and/or follow-up care. Elañe kwonaaj jorāān ilo ien eo kwoj bed ilo ekkatak in, jenaj jibañ eok kabbok jibañ eo kwoj aikuji. Ekoba first aid, jikin taktō ko rediñ, im jikin takto ko jet.

# What are the alternatives to being in this study?

#### Ta wāwein ko jet ijjelokin bed ilo ekkatak in?

You do not have to be in this study. Kwomaron jab bed ilo ekkatak in.

Organizations in the Republic of the Marshall Islands

PI (researcher): Sheldon Riklon, MD

■ There are no alternatives to being in this study, as it does not involve treatment or other procedures that may help you. Ejjelok bar jet wāwein ko jet nān bed ilo ekkatak in, einwōt an jab kōmman wāwein ko jet remaron jiban eok.

## Can I be taken out of the study even if I want to continue?

## Remaron ke kabojrak na jen ekkatak in elane ij konan wonmaanlok wot?

Yes, the study doctor (or head researcher) can take you out of the study if: Aet, taktō eo (ak eo ej bōk eddoin ekkatak in) remaron kabōjrak am bōk konaam ilo ekkatak in elañe:

- You do not follow study instructions. Kwojjab loori melele ko an ekkatak in.
- It is not in your best interest to continue. Ejjab ekkar im emman ñan kwe bwe kwon wonmaanlok wot.
- The study is stopped for any reason. Ekkatak in enaaj bojrak kon jabdrewot wun ko jejab maroñ ella joer.

#### What information will be collected about me in the study?

## Melele ta ko renaj būki jen na ilo ekkatak in?

During the study, we will need to learn private things about you, including Ilo ekkatak in, jenaj aikuj melele ko kōn kwe, einwōt

- General contact and background information about you, such as name, address, phone number, date of birth, sex, marital status and other demographic informationKilen topar eok im komeļeļe ko kon kwe, āinwot āt, atorej, talboon nomba, raan in ļotak, korā ak emmaan, mare, im meļeļe ko jet an juon jarlepju in arme
- Medical information about you, such as height, weight, pregnancy status, tests for diabetes, blood pressure, support from your family, managing your weight, exercise, and what you eat and drink Melele ko ikijien ājmour, einwōt joñan aitok, eddo, bōroro, kakōlkōl in tōñal, aibulat, jibañ jen baamle eo am, makūtkūt ak exercise, im mōñā ko kwoj kañi koba dren ko nimōm.
- If you are a patient of the RMI Ministry of Health and Human Services (MOHHS), we may request permission to get information about your diabetes care from your healthcare provider using your hospital patient number at 12 months after the end of the classes. Ne kwōj juon rinañinmej an RMI Ministry eo an Health im Human Services ak MOHHS, jemaron bok am mālim in kojerbal nomba in takto am ilo aujpitol nān bok meļeļe ikijien am takto in naninmej in tonal ilo naaj 12 allonālikin jemlokin kilaaj ko

Who will see this information? How will you keep it private?

Organizations in the Republic of the Marshall Islands

PI (researcher): Sheldon Riklon, MD

#### Won enaj loi melele kein? Ewi wawein am nej kojbaroki jen ro jet?

The local study team will know your name and have access to your information. Team eo loloodjake ekkatak in enej jelä etam im naaj loi melele ko am.

- We will do our best to make sure no one outside the study knows you are part of the study. Jenaj loloodjake im kōjbarok bwe ro rejjab bed ilo ekkatak in ren jab loi melele ko am.
- We will take your name off of information that we collect from you during the study.
  Jeban likit etam ilo melele ko am jenej buki jen kwe ilo ien ekkatak in
- When we share the results of the study in academic publications. We will not include your name or anything else that identifies you. Ne jenaj kwalok tobrak ko an ekkatak in ilo pepa ko an university ko, jeban likit etam ak jabdrewot melele ko renaj kallikar won kwe.
- If you chose to join the UAMS study Facebook group, other members in the group will know that you are participating in this research study. Access to the UAMS study Facebook page will be limited to enrolled participants and only the UAMS study staff serving as the administrator of the Facebook group will have permissions to add participants to the UAMS study Facebook group. You may still participate in the study even if you chose not to join the study Facebook group. Elañne kwar kālet in kobaļok ippān study Facebook group eo an UAMS, ro jet uwaan kurub eo renaaj jeļā ke kwōj bōk kuṇaaṃ ilo ekkatak in. Maron tōpar UAMS study Facebook peij eo enaaj nan wōt ro rej bōk kuṇaer im nan wōt rijerbal ro an ekkatak in an UAMS āinwōt administrator eo an Facebook group eo im ewor an mālim ko nan kadeļon ro rej bōk kwoṇaer ilo UAMS study Facebook group eo. Kwōj maron wōt bōk kuṇaaṃ ilo ekkatak in mene kwōj kālet in jab kobaļok ilo study Facebook group eo
- There are people who make sure the study is run the right way. These people may see information from the study about you. They are Ewor armij ro rej loloodjake bwe en jimwe an ettor ekkatak in. Armij rein remaron loi melele ko am. Armij rein rej
  - ✓ The research staff Rijerbal ro an ekkatak in,
  - ✓ OHRP (Office for Human Research Protections), a federal agency OHRP (Office for Human Research Protections), juon federal agency,
    - ✓ UAMS Institutional Review Board UAMS Institutional Review Board,
  - ✓ The Republic of the Marshall Islands Ministry of Health and Human Services Ministry eo an Health im Human Services eo an Republic eo an Marshall Islands,
    - ✓ Other institutional oversight offices Obiij ko rellaplok im rej etali jerbal kein,
- Ministry of Internal Affairs requires we tell the authorities if we learn Ministry eo an Internal Affairs ej aikuj bwe jen kōjeļāikļok ro tellokier eļanne jejeļā
  - about possible child or adult abuse K\u00f6n kakure ko \u00f1an ajiri ak rutto ro,

Organizations in the Republic of the Marshall Islands

PI (researcher): Sheldon Riklon, MD

that you might hurt yourself or someone else Elañe komaroñ kakure eok make ak ro jet,

## Where and how long will my information be kept?

### Melele ko aō renaj bed ia im ewi toon aer naj dābiji?

- We will code your information and keep the key to the code in a locked file. Kem naaj code ak nōmbaiki meļeļe ko am im likiti key nan code eo ilo juon bael eļak.
- Only designated research study staff will be able to link your information to you. Rijerbal ro wot rekkar ilo ekkatak in remaroñ jela nomba ta ko rej kallikar melele ko am.
- At the conclusion of the study, the data will be permanently de-identified and the key code will be destroyed. Ilo nej dedelok in ekkatak in, melele ko am naj jako im nomba ko nan melele ko am renej juloki.
- Your de-identified information will be destroyed seven years after the end of the research if you don't agree to let us keep your information for future research. Melele ko am renaj jako ālikin jiljilimjuon iiō ko ālikin an jemlok ekkatak in elañne kwonaj kwalok am jab kōnaan bwe jen kōjerbal melele ko am ñan ekkatak ko jet ilju im jeklaj

If I stop being in the study, what will happen to any information collected from me in the study? Elañe inaaj bōjrak jen ekkatak in, ta enaj walok ñan melele ko aō im emōj kar būki ilo ekkatak in?

• We will remove your data from the study if you tell us you want it removed. We will not be able to take your information out of the study after it has been published. Jenaaj kōmakit melele ko am jen ekkatak in elañe kwonaj ba jen jab kojerbali. Jejjab maron kōmakit melele ko am jen ekkatak in ālikin an mōj ad jeje pepa ikijien ekkatak in.

Will my information or samples from the study be used for anything else, including future research? Melele ko aō ak teej ko aō jen ekkatak in renaj ke kōjerbali nan jabdrewōt wāwein ko jet, koba nan ekkatak ko ilju im jōklaj?

- Yes. If you agree below, we will use the information in future research related to diabetes and other metabolic disease conducted by UAMS. Aet. Ne kwoj erra ijin ilal, kem naaj kojerbal meļele kein am ilo ekkatak ko an UAMS im renaaj kommani ilju im jekļaj im rej ekkejel ippan naninmej in tonal im naninmej ko jet rejelot wawein an anbwin ukwot mona im dren nan kajoor in ajmour.
  - O Personal identifiers will be removed and a special code or number with a key to the code will be kept separately. Information will be stored in a locked file, in a locked office consistent with UAMS policies. Electronic data will be in a password protected database with access restricted to research staff. Any paper documents containing your information will be assigned a unique identifying number and kept in a locked transfer case. If you change your mind about the use of your information in future

Organizations in the Republic of the Marshall Islands

PI (researcher): Sheldon Riklon, MD

studies, contact Dr. Sheldon Riklon at (479)713-8658. Melele ko rej kalikar won kwe kōmakiti im kojerbal nōmba ijelokin etam, im key eo nan nomba kein renaj kajenoloki. Melele ko renej kakuni ilo juon file emoj lake ekkar n̄an kakien ko an UAMS. Melele ko ilo computer ewōr aer password im ejjab aolep rijerbal ro an ekkatak in remaron̄ delon̄i. Jabdrewot pepa ko ewor melele ko am ie renaj kalikari kin juon am nomba, im laki ilo juon case ak kōbañ. Elan̄e kwonaj ukōt am lōmnak kōn kōjerbal melele kein am n̄an ekkatak ko iliju im joklaj, kūr lok Dr. Sheldon Riklon ilo (479)-713-8658.

- O Your information will not be shared with persons other than the current research staff. Jeban aji melele ko am ñan armij ro jet ijjelokin rijerbal ro ilo ekkatak in
- If you agree to let us keep your information for future research, we will keep it indefinitely. Elañe kwonaj errā bwe jen kōjerbal melele ko am ñan ekkatak ko ilju im jeklaj, innem melele ko am renaj bed wōt iumwin kōjparok ko an UAMS.
- If you don't agree to let us keep your information for future research, your information will be destroyed seven years after the end of the research. Elañe kwojjab errā bwe jen dābij melele ko am ñan ekkatak ko ilju im jeklaj, innem jenaj julok aolep melele ko am jiljimijuon iiō ālikin an jemlok ekkatak in.

# Will you tell me the results of the study?

Kom nej ke ba nan na kon tobrakin ekkatak in?

Yes. We will tell you and every person in the study about anything important that we discover from the study. Aet. Jenaaj kennanik eok im kajojo armij ro rej bed ilo ekkatak in kon jabdrewot melele ko reaurok renaj walok jen ekkatak in.

Will you tell me anything you learn that may impact my health?

#### Kom nej ke konnanok iio kon jabdewot wawein ko remaron jelet ajmour eo ao?

Yes. If we learn something about you that might be important for your health, we will tell you. Aet. Jenaaj konnanok eok elane enaaj walok jabdewot melele ko raurok ikijien ajmour eo am.

What if new information comes up about the study?

Ta enaaj walok elane ewor melele ko rokaal ikijien ekkatak in?

Organizations in the Republic of the Marshall Islands

PI (researcher): Sheldon Riklon, MD

We want you to know about anything that may change your mind about being in the study. Jōknaan bwe kwon jelā kon jabdewot melele ko im remaron jāniji am lomnak kon am bed ilo ekkatak in.

- The study team will let you know by: Team eo ej loloorjake ekkatak in enaaj konnaanik eok ilo an:
  - ✓ calling you call eok
  - ✓ sending you a letter jilkinwaj juon leta
  - ✓ telling you at a follow up visit kōnnanik eok ilo juon ian ien bar rool waj ko

# What if I have questions?

## Ak ne ewor ao kajjitok?

- Please call the local research team in the Marshall Islands at 692-456-4875, or the head researcher of the study Dr. Sheldon Riklon at (479)713-8658 or email at sriklon@uams.edu if you: Jouj im kūrļok local research team eo an Marshall Islands ilo 692-456-4875, ak rikappok meļeļe eo eutiej an ekkatak in Dr. Sheldon Riklon ilo (479)713-8658 ak email e ilo sriklon@uams.edu \_eļanne kwōj:
  - ✓ have any questions about this study ewor am kajjitōk ikijien ekkatak in,
  - ✓ feel you have been injured in any way by being in this study eñjake ke ewōr jorāān emōj an walok ilo am bed ilo ekkatak in
- You can also call the office at UAMS that supervises research if you can't reach the study team or want to speak to someone not directly involved with this study. To do so call the UAMS Institutional Review Board at 501-686-5667 during normal work hours. Komaron in tōbar rijerbal ro an UAMS ro rej loloorjake ekkatak in ne kwoj jab maron tōbar rijerbal ro ak kwoj kōnaan tōbar juon eo ejjab jerbal ilo ekkatak in. Kūr tok UAMS review board eo ilo 501-686-5667 ilo awa in jerbal ko.

Organizations in the Republic of the Marshall Islands

PI (researcher): Sheldon Riklon, MD

# University of Arkansas for Medical Sciences HIPAA Authorization Form

- Health Insurance Portability and Accountability Act of 1996 is the United States legislation that provides data privacy and security provisions for safeguarding medical information. Health Insurance Portability and Accountability Act of 1996 ej kakien eo an United States im ej kōmman kakien ko ikijien kōjbarok melele in taktō ko an armij
- The word "you" means both the person who takes part in the research, and the person who gives permission to be in the research. This form and the research consent form need to be kept together. Naan eo "kwe" ej jerbal ñan melele kein ruo: armij eo ej bōk konaan ilo ekkatak in koba armij eo ej letok mãlim in bed ilo ekkatak in. Pepa in koba pepa in mãlim eo (consent form) rej aikuj koba ibben dron ilo aer lewaj melele kein.

We are asking you to take part in the research described in the consent form. To do this research, we need to collect health information that identifies you. We may collect the following information: Jej kajitok bwe kwon bōk konaam ilo ekkatak in im emōj kōmeleleiki ilo pepa in consent form ak mālim eo. Ñan kōmmane ekkatak in, jenaj aikuj bōk melele ko rej kallikar wōn kwe. Jemaron naaj kajjitōk kōn melele kein:

- Hospital patient number nomba in takto
- date of birth raan in lotak
- sex kōrā/emmaan
- marital status emōj ke mare
- number of persons in your home jete armij ilo kabijuknen eo am
- education jikuul
- employment jerbal
- diabetes-related health conditions injuren
- insurance status naninmej ko jet remaron walok jen naninmej in tonal
- ability to access health care taktō
- race/ethnicity kwoj jen ia/lal eo am
- height aitokam
- weight eddoim
- pregnancy status bororo
- tests for diabetes kakōlkōl ko nan naninmij in tōnal
- tests for cholesterol kakölköl ko ñan nañinmij in kūriij
- blood pressure blood pressure ak aibōlat
- support from your family jiban jen baamle eo

Organizations in the Republic of the Marshall Islands

PI (researcher): Sheldon Riklon, MD

• managing your weight kojbarok am eddo

- exercise exercise ak makūtkūt
- Covid-19 vaccination history wā in COVID19 ko am
- what you eat and drink mona im dren ko nimom
- what medications you take uno ko kwōj būki

This information will be used for the purpose of learning more about teaching diabetes self-management. We will only collect information that is needed for the research. Participating in this research study will provide the following health information: Melele kein renaj kōjerbali ñan kōlablok melele ko ad ikkijien katak kin nañinmij in tônal im wāwein kōjbarok. Jenaaj bōk wōt melele ko jej aikuji ñan ekkatak in. Melele ko renaaj walok ilo am bōk konaam ilo ekkatak in rej einwōt:

- blood sugar levels jonan juka ak tonal eo ilo anbwinnum
- blood pressure levels jonan aer in botoktok ilo anbwinnum
- weight jonan eddo
- height jonan aitok
- BMI BMI ak jonan eddo eo ajmour im ekkar nan jonan am aitok

For you to be included in this research, we need your permission to collect, create and share this information. Bwe kwon bed ilo ekkatak in, kwoj aikuj letok mãlim bwe jen bõk melele ko am, kōbooji, im je pepa ko nan kwalok tōbrak in ekkatak in.

We will, or may, share your health information with people at the University of Arkansas for Medical Sciences (UAMS) who help with the research or things related to the research process, such as the study staff, the Republic of the Marshall Islands Ministry of Health and Human Services, the UAMS Institutional Review Board, and the research compliance office at the University of Arkansas for Medical Sciences. Kem naaj, ak maron, kwaļok meļeļe kon ājmour eo am ippān armej ro ilo University eo an Arkansas nan Medical Sciences ak UAMS me rej jipan tok ekkatak in ak wāwein ko rej ekkejel ippān wāwein jerbale ekkatak in, āinwot rijerbal ro an ekkatak in, Ministry eo an Health im Human Services eo an Republic eo an Marshall Islands, UAMS Institutional Review Board eo, im research compliance opiij eo ilo University eo an Arkansas nan Medical Sciences.

We may need to share your health information with people outside of UAMS who make sure we do the research properly, such as the Office for Human Research Protections and other institutional oversight offices. We believe that those involved with research understand the importance of preserving the confidentiality of your health information. However, some of the people outside of UAMS may share your health information with someone else. If they do, the same laws that UAMS must obey may not apply to others to protect your health information. Kom maron kwalok melele ko ikijien ajmour eo am ibben armij ro itulikin UAMS im rej loloorjake bwe en jimwe ad kommani ekkatak kein, einwot obiij eo an Office for Human

Organizations in the Republic of the Marshall Islands

PI (researcher): Sheldon Riklon, MD

Research Protections im obiij ko rej bar loloorjake ak koba lok ibbeir ilo aer jerbali kakien kein an ekkatak in. Jej kõtmene bwe ro rej bõk konaer ilo kõmmani ekkatak ko remelele aurõkin kõjbarok melele ko am. Bõtaab, jet armij ro itulikin in UAMS remaroñ lilok melele ko am ñan bar jet. Elañe renaaj, kakien eo UAMS ej aikuj loore remaroñ jab jelet er im remaroñ jab kõjbarok melele ko am.

This authorization to collect, use and share your health information expires at the end of the research study, unless you agree to allow us to use your de-identified information for future research at the bottom of this form. Mālim in nān ebbōk, kōjerbal im kwaļok meļeļe ko kōn ājmour eo am ej jemļok kitien ilo jemļokin ekkatak in, nān ne kwōj errā itulaļ in peba nān kōtļok am kōjerbal meļeļe ko am emoj joļok etam jen i nān ekkatak ko ilju im jekļaj.

If you sign this form, you are giving us permission to create, collect, use and share your health information as described in this form. You do not have to sign this form. However, if you decide not to sign this form, you cannot be in the research study. You need to sign this form and the research consent form if you want to be in the research study. Eļanīne kwōj jaini peba in, kwōj letok am mālim nān ejaak, ebbōk, kōjerbal im kwaļok meļeļe ko kōn ājmour ņe aṃ āinwōt an kōmeļeļe ilo peba in. Kwōjjab aikuj jaini peba in. Ijoke, eļanīne kwōj kālet in jab jaini peba in, kwōjjab nej maron pād ilo ekkatak in. Kwōj aikuj jaini peba in im peba in Mālim eo an ekkatak in eļanīne kwōj kōṇaan pād ilo ekkatak in.

If you sign this form but decide later that you no longer want us to collect or share your health information, you must either send a letter to Principal Investigator at the name and address below, or send an email to <a href="mailto:irb@uams.edu">irb@uams.edu</a>. Your letter or email must include: Eļanīne kwōj jaini peba in bōtaab kwokālet tokālik bwe ejako aṃ kōṇaan bwe kemin ebbōk ak kwaļok meļeļe kōn ājmour ņe aṃ, kwōj aikuj kōṇṇṇane juon iaan wāwein kein, jilkinļok juon leta nān eo ej bōk eddo in ebbōk meļeļe an ekkatak in ilo āt eo im atōrej eo ilaļ, ak jilkinļok juon email nān <a href="mailto:irb@uams.edu">irb@uams.edu</a>. Leta ak email eo aṃ ej aikuj kobaik:

- The study title (located at the top of this page) Taitol in ekkatak eo (ej pād itulon in peij in)
- A statement saying you changed your mind and are ending your "HIPAA Research Authorization" Juon ennaan ej ba bwe emoj am ukwot am lommak im kwoj kabojrak "HIPAA Research Authorization ak Komalim an Ekkatak eo an HIPAA"
- Your signature Am jain

You will need to leave the research study if we cannot collect and share any more health information. However, in order to maintain the reliability of the research, we may still use and share your information that was collected before the email or the Principal Investigator received your letter withdrawing the permissions granted under this authorization. Kwōnaaj aikuj in bōjrak jen ekkatak in eļañne kemij jab maron ebbōk im kwaļok elōnļok jabdewōt meļeļe ko kōn ājmour. Ijoke, nan dāpij wōt im kōjparok tiljek im mool eo an ekkatak in, kem maron wōt kōjerbal im kwaļok meļeļe ko am jekar būki mokta jen email eo ak an eo ej bōk eddo in ekkatak in loe leta in kabōjrak kōmālim ko am im rar kōmman iumwin kōmālim in.

Organizations in the Republic of the Marshall Islands

PI (researcher): Sheldon Riklon, MD

Etan Principal Investigator ak eo ej bōk eddo in ebbōk melele an ekkatak in:

Principal Investigator: Sheldon Riklon, M.D.

University of Arkansas for Medical Sciences Northwest

1125 North College Avenue Fayetteville, AR 72703 Telephone: (479) 713-8658

Email: sriklon@uams.edu

# By signing the document, I am saying:

# Ilo aō jaini pepa in, ij kallikar ke:

- ✓ I understand that joining this study is voluntary. Naij melele ke aō bebe bōk konaō ilo ekkatak in.
- ✓ I agree to be in the study. Naij errā in bed ilo ekkatak in.
- ✓ Someone talked with me about the information in this document and answered all my questions, uon armij ear konono ibba kon melele ko ilo pepa in im uwaaki aolep kajjitok ko aō.

#### I know that:

## Ijelā ke:

- ✓ I can stop any and all parts of the study at any time and nothing bad will happen to me. Imaron bojrak jabdewot ien ilo ekkatak in, im ejjelok joraan enaaj walok nan na.
- ✓ I can call or email the office that supervises research (UAMS Institutional Review Board) at 501-686-5667 or irb@uams.edu if I have any questions about the study or about my rights. I can also call 692-456-4875 or email wibing@uams.edu and speak with a member of the local research team in the Marshall Islands. Imaroñ kūr lok obiji eo ej bõk eddo in ekkatak ko (UAMS Institutional Review Board) ilo 501-686-5667 elañe ewōr jabdewōt kajjitōk ko ikijien ekkatak in ak ikijien maroñ ko aõ. Imaron bar kūrļok 692-456-4875 ak email e lok wibing@uams.edu im kenono ippān juon eo ej uwaan local research team eo ilo Marshall Islands.
- ✓ I do not give up any of my rights by signing this form. Ijjab julok maron ko aō ilo aō jaini pepa in.


| Study Title: Family Model of Diabetes Self-<br>Organizations in the Republic of Diabetes Self- | | -Management Education in Faith Based of the Marshall Islands |
|---|---|---|
| PI (researcher): | Sheldon Riklon, MD | |
| | | PID: |
| Laguas to be month | of this study. Noti anni in ha | d Slo obligatoly in |
| _ | of this study. Naij errā in be | a no ekkatak in |
| YES AET | □NO JAAB | |
| | k mālim bwe UAMS en kōjer | on from this study to other studies conducted bal melele ko aō ilo ekkatak ñan ekkatak ko |
| YES AET | NO JAAB | |
| conducted by UA im emōj joļok eta | MS in the Republic of the M | used for future diabetes related research<br>arshall Islands. Ij errā ñan an meļeļe ko aō<br>ekkatak ko an UAMS eo ilo Marshall Islands<br>l ippān nañinmej in tōñal. |
| YES AET | NO JAAB | |
| participant in thi | s study. Ij errā <b>nan an rijerb</b> | l short survey related to my experience as a al ro bar kūr tok ña ñan juon iien kajitōkin oi āinwōt juon eo ekar bōk kuṇaan ilo |
| YES AET | NO JAAB | |
| 0 | ontacted for future research<br>en ekkatak ko jet iliju im jōk | related to this study. Ij errā bwe ren<br>laj. |
| YES AET | NO JAAB | |
| Your name (please p | print) Etam (jouj im kallikare) | Your signature Jaini etam |
| Date Raan eo | | |
| | onsent name (please print) | Person Obtaining Consent signature |
| Armej eo ej bok mā | lim in (kallikar etam) | Jain eo an armej eo ej mālim in |

Date Raan eo